CLINICAL TRIAL: NCT00784680
Title: A Randomised, Double-Blind, Parallel Group Trial to Assess Quality of Life With Arimidex Alone, Nolvadex Alone, or Arimidex and Nolvadex in Combination, When Used as Adjuvant Treatment for Breast Cancer in Postmenopausal Women
Brief Title: ATAC - Quality of Life Sub-Protocol
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Francisco Sapunar, Medical Science Director, Arimidex and Faslodex, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 1033IE/0029; D5392C08389
Record Dates: First submitted 2008-11-03; First posted 2008-11-04 (Estimated); Last update posted 2009-05-01 (Estimated); Status verified 2009-04

CONDITIONS: Quality of Life
MeSH Terms: interventions — Anastrozole; Tamoxifen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Arimidex 1mg + Nolvadex placebo
  Interventions: Drug: Anastrozole
- 2 (Active Comparator): Arimidex placebo + Nolvadex 20mg
  Interventions: Drug: Anastrozole; Drug: Tamoxifen
- 3 (Active Comparator): Arimidex 1mg + Nolvadex 20mg
  Interventions: Drug: Tamoxifen

INTERVENTIONS:
Drug: Anastrozole — 1mg, orally, once daily
  Other Names: Arimidex
  Arms: 1; 2
Drug: Tamoxifen — 20mg, orally, once daily
  Other Names: Nolvadex
  Arms: 2; 3

SUMMARY:
To compare Quality of Life between the ARIMIDEX group, the NOLVADEX group and the ARIMIDEX plus NOLVADEX combination group during the first two years of treatment. (a) To compare the difference in Quality of Life between the ARIMIDEX group and the NOLVADEX group (b) To compare Quality of Life in the ARIMIDEX plus NOLVADEX combination group with the NOLVADEX group for non-inferiority; if non inferiority is concluded, the difference in QOL between these two groups will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for entry into the main ATAC trial 1033IL/0029
* Completion of a baseline questionnaire

Exclusion Criteria:

* Excluded from entry into the main ATAC trial (1033IL/0029)
* If, in the investigators opinion, the patient would be unable to comply with this sub-protocol due to psychiatric or literacy reasons

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 1998-04; Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Time to withdrawal
Time to recurrence